CLINICAL TRIAL: NCT06355271
Title: Quality of Postoperative Analgesia and Functional Recovery After Elective Cesarean Delivery Adding Different Doses of Intrathecal Fentanyl to Spinal Anesthesia With Bupivacaine and Intrathecal Morphine. A Single Center, Randomized, Multiple Blinded, Controlled Trial
Brief Title: Quality of Postoperative Analgesia and Functional Recovery After Elective Cesarean Delivery
Acronym: MoFe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Principal Investigator, Dossi Roberto, Dr. Med., Ente Ospedaliero Cantonale, Bellinzona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-00019
Record Dates: First submitted 2024-03-28; First posted 2024-04-09 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Obstetric Pain
Keywords: Cesarean section; Fentanyl; Functional Recovery
MeSH Terms: conditions — Labor Pain | interventions — 3-methylfentanyl

STUDY DESIGN:
Intervention Model Description: Single center, multiple-blind, prospective, randomized, controlled trial in 3 parallel groups
Who Masked: Participant, Care Provider, Investigator
Masking Description: Allocation will take place immediately before the intervention by the means of access to centralized, real-time allocation through a computer program. The identification code will be present on the data collection form (where the patient's name, surname or date of birth will not appear to ensure blinding of the study).
  Personnel not directly involved with patient care, present during the randomization process, will sterilely prepare anesthesia solution while maintaining a total volume of 3,1 ml. This will allow blinding of patients, care providers and data collectors. The procedure will take place as a common clinical practice in our center. When performing spinal anesthesia, sterility is of fundamental importance, so it will not be possible to have the syringe used tagged. In the kit all materials will be sterile
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Spinal anesthesia with no fentanyl
  Interventions: Procedure: Fentanyl 1
- Experimental 1 (Experimental): Spinal anesthesia with 10 mcg of fentanyl
  Interventions: Procedure: Fentanyl2
- Experimental 2 (Experimental): Spinal anesthesia with 20 mcg of fentanyl
  Interventions: Procedure: Fentanyl 3

INTERVENTIONS:
Procedure: Fentanyl 1 — Spinal anesthesia with a 27- gauge Whitacre needle at the L2-3 or L3-4 intervertebral space with the patient in sitting position with hyperbaric bupivacaine 0,5 %12 mg, 100 mcg of morphine, and no fentanyl
  Arms: Control
Procedure: Fentanyl2 — Spinal anesthesia with a 27- gauge Whitacre needle at the L2-3 or L3-4 intervertebral space with the patient in sitting position with hyperbaric bupivacaine 0,5 %12 mg, 100 mcg of morphine, and 10 mcg of of fentanyl
  Arms: Experimental 1
Procedure: Fentanyl 3 — Spinal anesthesia with a 27- gauge Whitacre needle at the L2-3 or L3-4 intervertebral space with the patient in sitting position with hyperbaric bupivacaine 0,5 %12 mg, 100 mcg of morphine, and 20 mcg of fentanyl
  Arms: Experimental 2

SUMMARY:
Based on randomization, patients will receive a mixture for spinal anesthesia and will be followed in the following hours for the various outcomes and for functional recovery

DETAILED DESCRIPTION:
In the study intervention group every patient will receive a spinal anesthesia composed by hyperbaric bupivacaine 12 mg 0,5 %, morphine sulfate 100 mcg and an added randomized dose of 10 or 20 mcg IT fentanyl. The spinal anesthetic will be administered with a 27 gauge Whitacre needle at the L2-3 or L3-4 intervertebral space with the patient in sitting position. Sterile saline will be used to dilute the mixture to a final volume of 3.1 mL. The allocated treatment will be kept a secret from the patient, the anesthesiologist managing the patient, and the entire study team. The fentanyl doses will be prepared by an anesthesiologist who will not be involved in the study or the patient's treatment. For 24 hours following surgery, each patient would receive intravenous patient-controlled morphine analgesia. In the control group every patient will receive a spinal anesthesia composed by hyperbaric bupivacaine 12 mg 0,5 % and morphine sulfate 100 mcg. The spinal anesthetic will be administered with a 27- gauge Whitacre needle at the L2-3 or L3-4 intervertebral space with the patient in sitting position. Sterile saline will be used to dilute the mixture to a final volume of 3.1 mL. The allocated treatment will be kept a secret from the patient, the anesthesiologist managing the patient, and the entire study team. For 24 hours following surgery, each patient would receive intravenous patient- controlled morphine analgesia.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 year of age
* height over 160 cm
* American Society Anesthesiologists physical status I and II
* term singleton parturients
* scheduled for elective cesarean delivery during spinal anesthesia at Ospedale Regionale Bellinzona Valli

Exclusion Criteria:

* patients with inability to consent
* patient refusal
* contraindication to spinal anesthesia (eg, hemodynamic instability, infection at the surgery site, and neurologic defects such as transverse myelitis)
* emergency cesarean delivery
* preeclampsia/eclampsia
* allergy to drugs used in the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — the study involves pregnant patients
Enrollment: 63 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Patient Controlled Analgesia morphine consumption | Day 1 after cesarean section
  Patient Controlled Analgesia morphine consumption in the first 24 postoperative hours
obstetric quality of recovery score | Day 1 after cesarean section
  obstetric quality of recovery score (ObsQoR-11)

SECONDARY OUTCOMES:
Visual Analogue Scale | Day 1 after cesarean section
  pain scores after surgery (Visual Analogue Scale -VAS- where 0 is the minimum value and 10 is the maximum value. The higher is the score the worse is pain control) at 4, 12 e 24 h.
pruritus | Day 1 after cesarean section (and day 0 for intraoperative pruritus)
  Intraoperative and postoperative pruritus (rating 0-10 The higher is the score the worse is pruritus)
nausea and vomiting; considering it as a dichotomous variable (yes or no), without evaluating its entity | Day 1 after cesarean section (and day 0 for intraoperative nausea and vomiting)
  intraoperative and postoperative nausea and vomiting
intraoperative hypotension | during the cesarean section
  intraoperative hypotension
intraoperative opioids | during the cesarean section
  intraoperative opioids in morphine equivalents
satisfaction rate | Day 1 after cesarean section
  satisfaction rate (0-100, where 0 is the minimum value and 100 is the maximum value. The higher is the score the better is the satisfaction rate)
intraoperative pain | during the surgery
  intraoperative pain Visual Analogue Scale (Visual Analogue Scale -VAS- where 0 is the minimum value and 10 is the maximum value. The higher is the score the worse is pain control)

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Regionale di Bellinzona, San Giovanni, Bellinzona, Switzerland

IPD SHARING:
Plan to Share IPD: No